CLINICAL TRIAL: NCT05316649
Title: Blood Loss Quantification During Major Abdominal Surgery: Study Protocol for a Prospective Cohort Trial.
Brief Title: Blood Loss Quantification During Major Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Defence, Faculty of Military Health Sciences (Other)
Collaborators: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Jan Zajak, Jan Zajak, MD, MA, University of Defence, Faculty of Military Health Sciences
Other Study IDs: BloodMO0FVZ0000503
Record Dates: First submitted 2022-03-20; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Blood Loss, Surgical; Blood Loss, Postoperative; Postoperative Complications
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Hemoglobin concentration Suctioned fluid Hemoglobin concentration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPB group: Adult patients undergoing for elective liver or pancreas surgery at Department of Surgery, University Hospital Hradec Kralove, Czech Republic.
  Interventions: Other: Measurement of external blood loss; Diagnostic Test: Serum Hemoglobin concentration

INTERVENTIONS:
Other: Measurement of external blood loss — Measurement of external blood loss
Diagnostic Test: Serum Hemoglobin concentration — Serum Hemoglobin concentration

SUMMARY:
Blood loss quantification during surgery remains unreliable and inaccurate. The purpose of the study is compare several methods of blood loss quantification in real surgical settings and to analyze the effect of blood loss on postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for liver or pancreatic surgery
* age of patient ≥ 18 years
* signed informed consent provided

Exclusion Criteria:

* patient coagulation disorder (congenital or iatrogenic due to the chronic use of anticoagulants).
* use of cell saver suctioning during operation
* damage/clotting of blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing for elective liver or pancreas surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood loos quantification | 1 year
  Estimated blood loss by surgeon (sEBL) Estimated blood loss by anesthesiologist (aEBL) Gravimetric blood loss weighted (vGBL) Calculated blood loos based on anthropometric and hematological parameters (vCBL) Spectrophotometric measured hemoglobin mass loss (hbMBL) Measured blood loss using using hbMBL and patient's average pre- and postoperative serum hemoglobin (vMBL)

SECONDARY OUTCOMES:
Postoperative complications | 1 year
  The effect of blood loss measured by spectrophotometric method on postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Zajak, MD, MA, Principal Investigator — University of Defence, Faculty of Military Health Sciences
Locations (1):
- University of Defence, Faculty of Military Health Sciences, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zajak J, Paral J, Sirovy M, Odlozilova S, Vinklerova K, Lochman P, Cecka F. Blood loss quantification during major abdominal surgery: prospective observational cohort study. BMC Surg. 2024 Jan 2;24(1):5. doi: 10.1186/s12893-023-02288-w. PMID 38166991